CLINICAL TRIAL: NCT07366190
Title: Effects of Premature Infant Oral Motor Intervention (PIOMI) on Feeding Behavior, Weight Gain, and Length of Hospital Stay in Preterm Infants: A Randomized Controlled Trial
Brief Title: PIOMI Effects on Preterm Infant Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Neslihan Altuntas Yilmaz, Principal Investigator, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEU-PT2025-04
Record Dates: First submitted 2025-12-15; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Prematurity
Keywords: Premature infant; PIOMI; breastfeeding behavior; weight gain; neonatal intensive care
MeSH Terms: conditions — Premature Birth; Weight Gain | interventions — Nursing Care

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment interventional model. Eligible preterm infants are randomly assigned to either the intervention group receiving Premature Infant Oral Motor Intervention (PIOMI) or to a control group receiving standard care. Both groups are followed concurrently throughout the study period, and outcome measures are assessed at baseline and after the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIOMI (Experimental): The PIBBS evaluates six sub-items: latching onto the breast, areola grasp, securing the breast with the mandible, sucking, longest sucking burst, and swallowing. Total scores were documented.
  In the intervention group, physiotherapists administered PIOMI, which consisted of cheek support, lip rounding, lip closure, gum massage, pressure on the lateral and anterior tip of the tongue, and palate tapping to stimulate sucking. The intervention lasted 3 minutes, followed by 2 minutes of non-nutritive sucking, administered twice daily for 7 consecutive days (each session lasting 5 minutes). Oxygen saturation and heart rate were monitored during the application.
  Interventions: Other: Premature Infant Oral Motor Intervention (PIOMI)
- Control (Other): The control group received routine nursing care without any additional oral motor stimulation.
  Interventions: Other: nursing care

INTERVENTIONS:
Other: Premature Infant Oral Motor Intervention (PIOMI) — The Beckman Oral Motor Intervention (BOMI) was redesigned by Dr. Brenda Lessen, modifying its duration and steps, to create the Premature Infant Oral Motor Intervention (PIOMI). PIOMI is the only preterm oral motor intervention that can be consistently and reliably applied and easily taught through a specific training program.In the intervention group, physiotherapists administered PIOMI, which consisted of cheek support, lip rounding, lip closure, gum massage, pressure on the lateral and anterior tip of the tongue, and palate tapping to stimulate sucking. The intervention lasted 3 minutes, followed by 2 minutes of non-nutritive sucking, administered twice daily for 7 consecutive days (each session lasting 5 minutes). Oxygen saturation and heart rate were monitored during the application.
  Arms: PIOMI
Other: nursing care — The control group received routine nursing care without any additional oral motor stimulation.
  Arms: Control

SUMMARY:
Objective: This study aimed to investigate the effects of Premature Infant Oral Motor Intervention (PIOMI) on body weight gain, breastfeeding behavior, and length of hospital stay in preterm infants hospitalized in the neonatal intensive care unit (NICU).

Methods: A randomized controlled experimental study design was used. A total of 32 preterm infants with gestational age between 26-30 weeks were randomly assigned to the intervention group (n=16) or control group (n=16). The intervention group received PIOMI twice daily for 7 consecutive days (14 sessions in total), while the control group received routine care only. The Premature Infant Breastfeeding Behavior Scale (PIBBS) was used to evaluate breastfeeding performance before and after the intervention. Weight changes and length of hospital stay were recorded and compared between groups.

DETAILED DESCRIPTION:
Objective

This study aimed to investigate the effects of Premature Infant Oral Motor Intervention (PIOMI) on feeding behavior, weight gain, and length of hospital stay in preterm infants hospitalized in the neonatal intensive care unit (NICU).

Methods

This study was designed as a randomized controlled experimental trial with a pretest-posttest parallel-group design. A total of 32 preterm infants with a gestational age between 26 and 30 weeks were randomly assigned to either the intervention group (n = 16) or the control group (n = 16). The intervention group received Premature Infant Oral Motor Intervention (PIOMI) twice daily for 7 consecutive days (14 sessions in total), while the control group received routine nursing care only. Breastfeeding behavior was assessed using the Premature Infant Breastfeeding Behavior Scale (PIBBS) before and after the intervention. Body weight was measured daily, and total weight gain and length of hospital stay were recorded. Statistical analyses were performed using appropriate parametric and non-parametric tests according to data distribution, with a significance level set at p < 0.05.

Conclusion

This study was designed to evaluate the clinical effects of PIOMI on feeding performance, weight gain, and hospitalization outcomes in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 26 and 30 weeks,
* Minimum birth weight of 1350 grams,
* Physical stability during oral stimulation,
* Apgar score of 4 or above at 5 minutes after birth.

Exclusion Criteria:

* Presence of congenital anomalies or chromosomal abnormalities,
* Chronic medical conditions such as bronchopulmonary dysplasia,
* Intraventricular hemorrhage (Grade III or IV),
* Necrotizing enterocolitis (NEC),
* Asphyxia and seizures,
* Treatments related to neonatal jaundice requiring exchange transfusion or blood transfusion,
* Sepsis confirmed by positive blood culture.

Ages: 24 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Premature Infant Breastfeeding Behavior Scale (PIBBS). | Baseline (pre-intervention) and Day 7 (post-intervention)
  The PIBBS evaluates six sub-items: latching onto the breast, areola grasp, securing the breast with the mandible, sucking, longest sucking burst, and swallowing. Total scores were documented.The Premature Infant Breastfeeding Behavior Scale (PIBBS) evaluates six sub-items: latching onto the breast, areola grasp, securing the breast with the mandible, sucking, longest sucking burst, and swallowing.
  The total score ranges from 0 to 20, with higher scores indicating better breastfeeding performance.
discharge weight | From baseline (pre-intervention) to day 7 after completion of the intervention
  Change in body weight from baseline to discharge
Length of Hospital Stay | From NICU admission (baseline) until hospital discharge, assessed up to 8 weeks
  Length of hospital stay is defined as the total number of days from admission to the neonatal intensive care unit (NICU) until hospital discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical restrictions and the vulnerable nature of the study population (preterm infants). Data contain sensitive clinical information, and sharing individual-level data could compromise participant confidentiality despite anonymization. Therefore, individual patient data will not be made publicly available.